CLINICAL TRIAL: NCT04413565
Title: Infection Rate of One-Stage Bilateral TKR - One Surgeon Sequential vs. Two Surgeon Simultaneous: A Randomized Controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Orkhan Aliyev, MD, Resident Doctor in Orthopaedic Surgery, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08.12.2016-71306642-050.01.04
Record Dates: First submitted 2020-05-29; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Infection Joint; Joint Infection; Arthroplasty Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two surgeon bilateral TKA group (Experimental): 2 surgeons will perform simultaneous total knee arthroplasty in this group.
  Interventions: Procedure: Simultaneous bilateral total knee arthroplasty
- Single surgeon bilateral TKA group (Active Comparator): One surgeon will perform sequentially tptal knee arthroplasty in this group
  Interventions: Procedure: Sequenced bilateral TKA

INTERVENTIONS:
Procedure: Simultaneous bilateral total knee arthroplasty — Two surgeon bilateral TKA group
  Arms: Two surgeon bilateral TKA group
Procedure: Sequenced bilateral TKA — Single surgeon bilateral TKA group
  Arms: Single surgeon bilateral TKA group

SUMMARY:
The use of bilateral total knee replacements (TKR) is increasing with the number of patients with bilateral end-stage knee osteoarthritis. Bilateral TKR can be performed in three different ways: single-stage, two-team simultaneous bilateral TKR (two surgeons bilateral TKR); single-stage, a sequential bilateral TKR (single surgeon bilateral TKR); and two-stage bilateral TKR. Periprosthetic joint (PJI) infections are serious complications after TKR that negatively affect the aimed outcome, decrease patient satisfaction, and increase morbidity and mortality. The incidence of PJI is 1-2% and the number of cases is projected to grow as the indications for TKR continue to increase. Investigators will prospectively compare the incidence of periprosthetic joint infection between groups.

DETAILED DESCRIPTION:
924 knees (462 participants) will prospectively be randomized into 2 groups: two surgeons bilateral TKA and single surgeon bilateral TKA. While 2 surgeons will perform simultaneous total knee arthroplasty in the two surgeons' bilateral TKA group, one surgeon will perform sequentially in the single surgeon bilateral TKA group. The primary outcome is to compare the incidence of PJI between the groups. Secondary, logistic regression use to estimate the effect of two surgeons bilateral TKA and single surgeon bilateral TKA on the likelihood of a patient being infected.

ELIGIBILITY:
Inclusion Criteria:

Primary bilateral knee osteoarthritis with refractory to conservative treatment Patients who accept participation in the research and the randomization

Exclusion Criteria:

no history of malignancy without severe extra-articular deformities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Estimated)
Dates: Start 2016-12-08 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Infection incedence | 90 days
  Early infection rates

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No